CLINICAL TRIAL: NCT02601534
Title: Be Healthy, So Easy: FAMILY Education Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Caritas Medical Centre, Hong Kong (Other); The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Project Manager (Health Communication), The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UW 15-330
Record Dates: First submitted 2015-11-05; First posted 2015-11-10 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Hypokinesia
Keywords: sedentary behaviour; physical activity
MeSH Terms: conditions — Hypokinesia; Motor Activity | interventions — Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zero-time Exercise (PA) group (Experimental): The intervention arm (PA group) aims to improve family communication and well-being, reduce sedentary behavior and increase physical activity. The programme includes a knowledge and motivation enhancement session at baseline, an experience sharing session at 3 months, a family gathering session at 6 months, and a holistic health session at 12 months after the first session as well as biweekly/monthly mobile messages.
  The holistic health session is not a part of the cRCT, it aims to collect one-year feedback from participants and provides additional health information to improve dietary habits.
  Interventions: Behavioral: Zero-time Exercise
- Healthy Eating (HE) group (Placebo Comparator): The control arm (HE group) aims to improve family communication and well-being and enhance healthy eating habits. Participants are required to engage their family members in their activities. The programme includes a knowledge and motivation enhancement session at baseline, an experience sharing session at 3 months, a family gathering session at 6 months, and a holistic health session at 12 months after the first session as well as biweekly/monthly mobile messages.
  The holistic health session is not a part of the cRCT, it aims to collect one-year feedback from participants and provides additional health information to improve physical activity habit.
  Interventions: Behavioral: Healthy Eating

INTERVENTIONS:
Behavioral: Zero-time Exercise — a knowledge and motivation enhancement session at baseline, an experience sharing session at 3 months, a family gathering session at 6 months, and a holistic health session at 12 months (not a part of cRCT, for the collection of feedback only) as well as biweekly/monthly mobile messages to improve physical activity habit.
  Arms: Zero-time Exercise (PA) group
Behavioral: Healthy Eating — a knowledge and motivation enhancement session at baseline, an experience sharing session at 3 months, a family gathering session at 6 months, and a holistic health session at 12 months (not a part of cRCT, for the collection of feedback only) as well as biweekly/monthly mobile messages to improve dietary habit.
  Arms: Healthy Eating (HE) group

SUMMARY:
The goal of the study is to evaluate the effectiveness of a family-focused, interactive, and theory-based intervention to reduce the sedentary behavior and increase physical activity, family communication and well-being of the participants.

The intervention is to use Zero-time Exercise, the positive psychology theme "Appreciation and Gratitude" [23, 24], and role modelling approach to get sedentary people to start exercising, increase levels of physical activity, family communication and well-being of the participants and their family members.

The intervention aims to encourage positive and sustainable health actions among participants and their family members.

DETAILED DESCRIPTION:
Lack of physical activity is a behavioural risk for non-communicable diseases. The World Health Organization (WHO) reported that physical inactivity and unhealthy diets are two of the four main behavioural risk factors that contribute to non-communicable diseases. Globally, people who are overweight and obese, particularly if these people are physically inactive. They are at risk for morbidity and mortality.

Hong Kong-specific data demonstrates that many people cannot meet World Health Organization targets for physical activity. The Hong Kong Behavioural Risk Factor Survey reported that, for the seven days prior to the survey, about half (52.0%) of adults aged 18-64 had not done any moderate physical activity. Overall, only 37.5% of the respondents met the WHO's recommended physical activity level of at least 150 minutes of moderate or 75 minutes of vigorous physical activity a week for adults.

There is emerging evidence of effective behavioral interventions to decrease sedentary behavior. Some studies focused on reducing screen time or active workstations that encourage standing at the computer. Others focus on increased use of stairs instead of lifts. These interventions used behaviour change techniques such as goal-setting and behavioural self-monitoring. As previous approaches have not shown promising results, new approaches are needed to reduce sedentary behaviour and increase exercise or physical activity.

The goal of the study is to evaluate the effectiveness of a family-focused, interactive, and theory-based intervention to reduce the sedentary behavior and increase physical activity of the participants.

The intervention is to use Zero-time Exercise, the positive psychology theme "Appreciation and Gratitude", and role modelling approach to get sedentary people to start exercising, increase levels of physical activity, family communication and well-being of the participants and their family members. The intervention aims to encourage positive and sustainable health actions among participants and their family members.

Needs assessment and focus group interview will be conducted before program design and after conducting the training, respectively. Process evaluation will be performed to evaluate the process of each component of the program. Qualitative and quantitative assessments will be used to evaluate the effectiveness of this Zero-time Exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Parents with at least on child between 3 and 18;
2. Parents with at least primary school educational level:
3. Parents who can read and write Chinese.

Exclusion Criteria:

1. People with a serious health condition that might prevent them from participating in physical activity;
2. Parents who do not have a child between 3 and 18.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 673 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in behavior on performing physical activity in relation to Zero-time Exercise, moderate and vigorous exercises | baseline, 3 months
  Behaviors on performing physical activity will be assessed by outcome-based questionnaire

SECONDARY OUTCOMES:
Change in behavior on performing physical activity in relation to Zero-time Exercise, moderate and vigorous exercises | baseline, 3 months, 6 months, 1 year
  Behavior on performing physical activity will be assessed by outcome-based and physical activity questionnaire
Change in behavior on taking healthy diet | baseline, 3 months, 6 months, 1 year
  Behavior on taking healthy diet will be assessed by outcome-based healthy diet questionnaire
Attitude on performing Zero-time Exercise, | immediate after training session, 3 months, 6 months, 1 year
  Attitude on performing physical activity in relation to Zero-time Exercise will be assessed by outcome-based questionnaire
Perceived ability and intention to motivate participants themselves and their family to increase Zero-time Exercise | baseline, 3 months, 6 months, 1 year
  Perceived ability and intention to motivate participants themselves and their family members on performing Zero-time Exercise will be assessed by outcome-based questionnaire
Change in participants' own health and happiness | baseline, 3 months, 6 months, 1 year
  Personal health and happiness will be assessed by outcome-based questionnaire
Change in participants' family harmony | baseline, 3 months, 6 months, 1 year
  Family harmony will be assessed by outcome-based questionnaire
Change in physical fitness performance (Endurance) | baseline, 3 months,6 months, 1 year
  Endurance will be assessed through a simple fitness test called foot pedaling
Family members' behavior on performing physical activity in relation to Zero-time Exercise, | 6 months
  Family members' behavior on performing physical activity in relation to Zero-time Exercise will be assessed by outcome-based questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK Lai, DN, Principal Investigator — The University of Hong Kong
Locations (1):
- Caritas integrated Family Service Centre, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Lai AYK, Lam EYW, Fabrizo C, Lee DPK, Wan ANT, Tsang JSY, Ho LM, Stewart SM, Lam TH. A Community-Based Lifestyle-Integrated Physical Activity Intervention to Enhance Physical Activity, Positive Family Communication, and Perceived Health in Deprived Families: A Cluster Randomized Controlled Trial. Front Public Health. 2020 Sep 15;8:434. doi: 10.3389/fpubh.2020.00434. eCollection 2020. PMID 33042934
- See also: World Health Organization (2017). Noncommunicable diseases : Fact Sheet — http://www.who.int/en/news-room/fact-sheets/detail/noncommunicable-diseases
- See also: Department of Health (2016). Behavioural Risk Factor Survey — https://www.chp.gov.hk/files/pdf/brfa_report_april_2016_eng.pdf